CLINICAL TRIAL: NCT01458756
Title: Evaluation of Psychological Defense Mechanisms Used by Liver Transplant Patients on Their Somatic Psychological and Social Outcome. Research for Protective or Vulnerability Factors.
Brief Title: Study of Psychological Defense Mechanisms Used by Liver Transplant Patients
Acronym: GHEPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2006_0623; DGS 2006/0393 (Other: AFSSAPS)
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Liver Diseases
Keywords: liver transplant patients; hepatic transplantation
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver transplant patients: Population of adult patients awaiting liver transplant, status on the waiting list in the transplant center of University Hospital of Lille.

SUMMARY:
Organ transplantation has a special place in the medical field. It symbolizes a medicine whose limits always seem to be repelled. Because transplantation is unusual, it places people in front of outstanding issues which he has to cope with his personality and history. Factors involved in the psychology of patient presenting with graft are past and present psychic functioning, object relations, experience of transplantation itself and quality of social environment.

Before or after graft defense mechanisms can be so intense that they can make the patient unable to overcome the graft. Yet as a pathological mechanism that denial was considered beneficial provided it is short.

The aim of this study is to evaluate on psychopathological influence of psychological defense mechanisms used by liver transplant patients on their somatic psychological and social outcome.

DETAILED DESCRIPTION:
The objective is to measure the influence of variations of psychological defense mechanisms.

The investigators want to measure the influence of personal history of patients, causal disease pre-existing, conditions of graft's realization, structure of patient's social environment (family or institutional); and wish to identify which of those elements can be protective or vulnerability factors with a view to allow adequate support (especially for patients who had multiple poor prognostic factors)

The investigators will study pre-transplant psychological defense mechanisms of the subjects using the Bond Defense Style Questionnaire and structure of personality using the SCID II personality scale. They will evaluate post-transplant patient outcomes on clinical and social developments with DSQ 88 and General Health Questionnaire (GHQ 28) to six months, twelve months and five years after transplantation. Meanwhile, they will address each time you visit the data on consumption, misuse and alcohol dependence using the AUDIT questionnaire (Alcohol Use Disorders Identification Test).

The hypothesis is that the defense mechanisms, their variations and personality of the patients are both vulnerability factors as protective factors in different phases of the graft. Identification should allow to optimize care and improve overall health. Results of this research could make it possible to determine the factors used in liaison psychiatry in the long term to ensure an adequate medical and psychiatric support to transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients between 18 and 65 years old
* liver disease requiring a liver transplantation
* registered on the waiting transplant list in the University Hospital of Lille

Exclusion Criteria:

* fulminant hepatitis
* mental incapacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients awaiting liver transplantation and registered on the waiting list in the transplant center of University Hospital of Lille
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2006-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change in Bond Defense Style Questionnaire 88 | baseline and 6 months and 1 year and 5 years
  Change in psychological defense mechanisms measured by the Defense Style Questionnaire 88, prior and after liver transplantation

SECONDARY OUTCOMES:
personality disorders evaluation by SCID II personality scale | baseline and 6 months and 1 year and 5 years
  structure of personality using the SCID II personality scale
Minimal International Neuropsychiatric Interview MINI results | 6 months and 1 year and 5 years
  presence of psychopathological disorders evaluated by MINI six months, one year and five years after liver transplantation
Alcohol Use Disorders Identification Test AUDIT score | baseline and 6 months and 1 year and 5 years
  consumption, misuse and alcohol dependence measured by AUDIT score
Change in mental health level by General Health Questionnaire GHQ 28 | baseline and 6 months and 1 year and 5 years
  Change in mental health levl measured by the General Health Questionnaire GHQ 28, prior and after liver transplantation
social evolution | baseline and 6 months and 1 year and 5 years
  change in professional, family , financial states

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, Lille, France